CLINICAL TRIAL: NCT00270387
Title: Prospective Randomized Outcomes Study of Acutely Decompensated Congestive Heart Failure Treated Initially in Outpatients With Natrecor (Nesiritide) - The PROACTION Trial
Brief Title: A Study of Short-Term Outcomes and Economic Impact For Patients With Worsening Congestive Heart Failure When Natrecor (Nesiritide) is Added to Standard-Care Therapy, Compared to Administration of Placebo With Standard-Care Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005209
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Cardiomyopathies; Heart Failure, Congestive; Dyspnea, Paroxysma
Keywords: Acutely Decompensated Congestive Heart Failure; Heart Failure; Renal Impairment; Kidney Failure; Myocardial Infarction.
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Dyspnea; Renal Insufficiency; Myocardial Infarction | interventions — Natriuretic Peptide, Brain

ARMS (1):
- 001 (Experimental): Natrecor (nesiritide)
  Interventions: Drug: Natrecor (nesiritide)

INTERVENTIONS:
Drug: Natrecor (nesiritide)

SUMMARY:
The purpose of this pilot study is to compare the clinical effects, safety profile, and economic impact of standard therapy plus NatrecorÂ® (nesiritide, a recombinant form of the natural human peptide normally secreted by the heart in response to heart failure) to standard therapy plus placebo in patients who present to the Emergency Department with worsening congestive heart failure (CHF) and are treated in the Emergency Department /Observation Unit.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) is a public health epidemic in the U.S., affecting almost 5 million Americans. It is associated with a 5-year mortality rate of 50% (according to the American Heart Association, 1999) and is currently the most costly cardiovascular disease in the U.S. (according to Rich MW et al 1999 and O'Connell JB 2000). In 1999, the total estimated direct and indirect costs associated with the treatment of CHF approached $56 billion (according to O'Connell JB 2000). Advanced CHF accounts for over 1 million hospital admissions annually in the U.S.and for a large portion of the total expense to third-party payers, due to the high cost of acute inpatient care and related Emergency Department visits.

Emergency Departments are the last line of defense against hospital admission for CHF. Operational and liability issues that pertain to the typical Emergency Department lead to hospital admission for most CHF patients. Yet, problems with bed availability may lead to the delayed transfer of patients from the Emergency Department to the inpatient unit, further delaying important treatment. To address this, many Emergency Departments have developed extended-stay policies for the observation and continuing care of patients who cannot be discharged from the Emergency Department within a few hours of arrival. With an extended stay (< 24 hours) for evaluation and treatment in the Emergency Department, hospital admission for CHF may be significantly reduced by adequately ruling out coronary ischemia and aggressively treating the precipitating factor of the decompensation. This allows physicians to better assess the appropriateness of admission for the patient (according to Graff LG 1993 ). Initiation of a safe and effective acute therapy in addition to usual standard care may make it possible to further reduce hospital admissions or the severity of the patient's condition at the time of the admission.

Natrecor® has been approved for use in the treatment of acutely decompensated CHF patients with dyspnea at rest or with minimal activity. It is a recombinant form (produced by genetic engineering) of naturally occurring human B-type natriuretic peptide (BNP, also known as brain natriuretic peptide) produced primarily by the ventricular myocardium (according to Hosoda K et al 1991). Natrecor® has been well tolerated in controlled clinical trials involving more than 1000 patients with CHF. The data from these previous studies suggest that doses of Natrecor® may be a potent agent for the treatment of acute CHF with a unique combination of desirable effects on the flow of blood throughout the body; the hormones secreted by the nervous system; and support of copious salt outputs by the renal system not provided by currently available therapies (according to LeJemtel TH et al 1998). Although Natrecor® has not been studied in the setting of an Emergency Department, it has been administered as a fixed-dose infusion without invasive monitoring to over 500 patients. Furthermore, Natrecor® has not been associated with an increase in cardiac ectopy or arrhythmias in both placebo-controlled and active-controlled trials (according to Burger AJ et al 1999 and Mills RM et al 1999).

This multicenter, randomized, double-blinded pilot study compares the clinical effects, safety profile, and economic impact of standard therapy plus Natrecor® to standard therapy plus placebo in the treatment of acutely decompensated CHF in an Emergency Department/Observation Unit setting. Study drug (Natrecor® or placebo) is administered as a bolus of 2 mcg/kg over approximately 60 seconds, immediately followed by a fixed-rate infusion of 0.01 mcg/kg/min for at least 12 hours. Subjects who continue to receive study drug and who remain in the Emergency Department/Observation Unit beyond 12 hours, up to 24 hours, have vital signs measured at 18 hours, 24 hours, immediately before discontinuation of study drug, and at 30 minutes, 1 hour, and 2 hours after discontinuation of study drug. Also, global clinical and dyspnea (difficulty breathing and shortness of breath) evaluations, and a visual monitoring scale for dyspnea, are completed at the time of termination of study drug in the Emergency Department/Observation Unit, or admission to the hospital. The health-economic analysis focuses on resource utilization and cost of care for initial treatment in the Emergency Department/Observation Unit and inpatient facility (if admitted), as well as any subsequent treatment in an Emergency Department or acute inpatient facility within the 30-day study period.

The study hypothesis is that the efficacy and safety profile of Natrecor® may be conducive to its early administration for acute treatment of heart failure in the Emergency Department and that in addition to standard care, may make it possible to further reduce hospital admissions or the severity of the patient's condition at the time of admission. Natrecor® 1.5 mg for injection made up to final concentration of 0.3 mg/mL with 5% dextrose in water, or placebo. Dispensed as an intravenous bolus of 2 mcg/kg over approximately 60 seconds, immediately followed by a fixed-rate infusion of 0.01 mcg/kg/min for at least 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history consistent with congestive heart failure (either chronic or new onset) with fluid overload or elevated cardiac filling pressures by clinical diagnosis
* having a need for observation and intravenous therapy for at least 12 hours, primarily for the treatment of acutely worsening heart failure
* having dyspnea (difficulty breathing and shortness of breath) at rest, while supine, or immediately upon minimal exertion, and evidence of heart failure rather than pulmonary disease as the primary cause for the dyspnea
* having jugular venous distension, abdominal discomfort (such as decreased appetite or nausea) and a weight gain of at least 5 pounds in the previous month
* having chest x-ray findings indicative of heart failure, or rales (sounds associated with fluid in the lung cavity) heard on physical examination.

Exclusion Criteria:

* Patients having a clinical status so acutely unstable that invasive monitoring or mechanical ventilation is required
* admitted to Emergency Department/Observation Unit primarily for a diagnostic evaluation (such as ruling out myocardial infarction or to diagnose irregular heart beats)
* having systolic blood pressure consistently less than 90 mm Hg
* having cardiogenic shock (a sudden decrease in blood pressure that results in decreased perfusion of body tissues and organs), volume depletion, or any other clinical condition that would contraindicate the administration of intravenous diuretics, ACE inhibitors, or an intravenous agent with potent vasodilating properties
* having a circumstance recognized at baseline evaluation that would definitely prohibit discharge to home from the Emergency Department/Observation Unit in less than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2001-01; Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Natrecor® can be safely administered in outpatient settings with blood pressure monitoring; Number of hospital readmissions and average length of stay in the hospital

SECONDARY OUTCOMES:
Economic Impact on hospitals of earlier and more aggressive treatment in the Emergency Department with Natrecor® added to standard care

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- [Result] Peacock WF 4th, Holland R, Gyarmathy R, Dunbar L, Klapholz M, Horton DP, de Lissovoy G, Emerman CL. Observation unit treatment of heart failure with nesiritide: results from the proaction trial. J Emerg Med. 2005 Oct;29(3):243-52. doi: 10.1016/j.jemermed.2005.01.024. PMID 16183441
- See also: SCIOS Submits Interim Report to FDA — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=967&filename=CR005209_CSR.pdf